CLINICAL TRIAL: NCT05754710
Title: Korean Post-marketing Surveillance for Xeljanz® 5 mg Film-coated Tablets and Xeljanz® 1 mg/mL Oral Solution in Patients With Active pJIA and jPsA
Brief Title: Korea Xeljanz Post-marketing Surveillance for Juvenile Idiopathic Arthritis
Acronym: KRXeljanzJIA
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921400; Xeljanz JIA PMS (Other: Alias Study Number)
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis, Juvenile; Polyarticular Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Drug: Xeljanz — Juvenile Idiopathic Arthritis (JIA) patients with Xeljanz

SUMMARY:
This study is to assess the safety and effectiveness of Xeljanz in Juvenile Idiopathic Arthritis (JIA) patients in routine clinical practice in Korea. JIA patients experience persistent joint pain, swelling and stiffness. This is a prospective observational study.

Xeljanz is a JAK inhibitor. It was first approved in 2014 for rheumatoid arthritis patients in Korea. The ministry of Food and Drug Safety in Korea mandates for a drug manufacturer to report the post-marketing surveillance after drug's approval or indication extension. This study is to see the safety and effectiveness of Xeljanz in Juvenile Idiopathic Arthritis patients in routine clinical practice in Korea.

This study is seeking patients who:

* Are 2 to less than 18 years of age;
* Are given Xeljanz for the treatment of JIA.

The study sponsor will monitor patients' treatment experience for up to 44 weeks. This will help assess the safety and effects of this study medicine.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Pediatric subjects aged from 2 years to less than 18 years
2. Xeljanz administered according to efficacy/effectiveness on the approved labeling
3. Patients who will administer Xeljanz based on the medical judgement of the investigator
4. Evidence of a personally signed and dated informed consent document indicating that the subject (and a legally acceptable representative) has been informed of all pertinent aspects of the study

Exclusion Criteria:

Subjects meeting any of the following criteria will not be included in the study:

1) Subjects who are contraindicated from taking Xeljanz according to approved labeling*

*Refer to most recently approved label

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with active polyarticular Juvenile Idiopathic Arthritis or juvenile Psoriatic Arthritis who are administered Xeljanz according to the approved label in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment emergent treatment-related adverse events | Maximum of 12 months from the time of first administration of Xeljanz
  Incidence of each adverse event (AE) will be presented with 95% confidence interval. Serious, related, and/or unexpected AEs will be summarized separately. Additionally, in the event that AEs designated as important potential risks and important identified risks are reported, or if a patient in the missing information group is recruited, related safety information will be provided separately.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921400